CLINICAL TRIAL: NCT03911063
Title: A Single-Blind Placebo-Controlled Telemedicine Clinical Trial for Cognitive Behavioral Therapy in Familial Dysautonomia
Brief Title: Telemedicine Clinical Trial for Cognitive Behavioral Therapy in Familial Dysautonomia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Personnel unavailable to run the study
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-01152
Record Dates: First submitted 2019-03-28; First posted 2019-04-10 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Familial Dysautonomia
Keywords: Telemedicine
MeSH Terms: conditions — Dysautonomia, Familial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral therapy (CBT) (Experimental)
  Interventions: Behavioral: CBT sessions
- Placebo Talking Sessions (Active Comparator)
  Interventions: Behavioral: Talking Sessions

INTERVENTIONS:
Behavioral: CBT sessions — weekly 20-40 min CBT sessions during 8 weeks; Both the talking sessions (i.e., placebo) and CBT sessions will be performed via telemedicine either via a HIPAA secure telemedicine platform or the telephone based on the preference of the individual patient.
  Arms: Cognitive behavioral therapy (CBT)
Behavioral: Talking Sessions — 20-40 min talking sessions (i.e., placebo) for 8 weeks; The placebo talking sessions will be performed by an acute care and palliative care board certified, New York State licensed nurse practitioner at the NYU Dysautonomia Center who is familiar with each FD subject enrolling in the study and an expert in familial dysautonomia. The NP will focus the 20-40 minute conversation on typical medical questions and concerns that the FD patient routinely calls the Center to discuss.
  Arms: Placebo Talking Sessions

SUMMARY:
This is a single-blind, placebo-controlled, telemedicine clinical trial to assess the efficacy of cognitive behavioral therapy (CBT) in adult patients 18 years and older with familial dysautonomia (FD) and anxiety and/or depression and/or obsessive compulsive or related disorders. The trial will enroll 20 adult patients each with FD who have anxiety and/or depression and/or obsessive compulsive or related disorders by the DSM V criteria.

Enrolled participants will be allocated to receive, in a non-randomized fashion, weekly 5-10 min talking sessions (i.e., placebo) for 8 weeks, followed by weekly 30-60 min CBT sessions during 8 weeks. Although investigators will be un-blinded to the intervention, participants will be blinded to the expected effects of each intervention.

Both the talking sessions (i.e., placebo) and CBT sessions will be performed via telemedicine either via a HIPAA secure telemedicine platform or the telephone based on the preference of the individual patient. If a patient specifically requests talking or CBT sessions to be performed in person, this will be accommodated. The use of telemedicine is to accommodate disability and potential physical limitations of this unique patient population. The CBT sessions will be supervised by Lily Armstrong, certified mental health therapist and Dr. Thomas Boes, NYU Clinical Assistant Professor in the Departments of Psychiatric and Neurology.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of familial dysautonomia (FD).
* DSM-V criteria of major depressive disorder OR anxiety disorder OR obsessive-compulsive behaviors.
* STAI score ≥ 25 OR a PHQ-9 depression scale score ≥ 5 or greater.
* Willing and able to complete 8 sessions of placebo and 8 sessions of CBT.
* If taking an antidepressant it will be maintained at a constant dose throughout study and concurrent talk therapy from another therapist will not be initiated during the study.
* MoCA score of 14 or greater.

Exclusion Criteria:

* Current suicidal attempt or suicidal ideation (subjects with a past history of suicidal ideation or attempt are eligible to participate).
* Patients starting psychoactive medications within 3-months prior to screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
STAI anxiety score | Baseline
  The range of possible scores for form Y of the STAI varies from a minimum score of 20 to a maximum score of 80 on both the STAI-T and STAI-S subscales. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
STAI anxiety score | Week 2
  The range of possible scores for form Y of the STAI varies from a minimum score of 20 to a maximum score of 80 on both the STAI-T and STAI-S subscales. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
STAI anxiety score | Week 9
  The range of possible scores for form Y of the STAI varies from a minimum score of 20 to a maximum score of 80 on both the STAI-T and STAI-S subscales. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
STAI anxiety score | Week 17
  The range of possible scores for form Y of the STAI varies from a minimum score of 20 to a maximum score of 80 on both the STAI-T and STAI-S subscales. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
PHQ-9 depression score | Baseline
  9 item depression scale of the patient health questionnaire.The total sum of the responses suggests varying levels of depression. Scores range from 0 to 27. In general, a total of 10 or above is suggestive of the presence of depression.
PHQ-9 depression score | Week 2
  9 item depression scale of the patient health questionnaire.The total sum of the responses suggests varying levels of depression. Scores range from 0 to 27. In general, a total of 10 or above is suggestive of the presence of depression.
PHQ-9 depression score | Week 9
  9 item depression scale of the patient health questionnaire.The total sum of the responses suggests varying levels of depression. Scores range from 0 to 27. In general, a total of 10 or above is suggestive of the presence of depression.
PHQ-9 depression score | Week 17
  9 item depression scale of the patient health questionnaire.The total sum of the responses suggests varying levels of depression. Scores range from 0 to 27. In general, a total of 10 or above is suggestive of the presence of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Kaufmann, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States